CLINICAL TRIAL: NCT02438969
Title: (Epi)Genetic Modulators of Fear Extinction in Alcohol Dependence
Brief Title: Epi-Genetic Modulators of Fear Extinction in Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150127; 15-AA-0127
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-03-10

CONDITIONS: Fear; Stress; Alcohol Dependence
Keywords: Alcohol; Alcohol Dependence; Stress; Fear Conditioning; Natural History
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (4):
- AUD/ELS-: Treatment seeking or non-treatment seeking individuals with AUD without ELS exposure
- AUD/ELS+: Treatment-seeking or non-treatment seeking individuals with AUD and early life stress (ELS) exposure
- non-AUD/ELS-: non-AUD controls without ELS exposure
- non-AUD/ELS+: Non-AUD controls with ELS exposure

SUMMARY:
Background:

- Researchers want to learn if people with alcohol dependence have more difficulty learning to feel calm, or learn to fear things more easily. They also want to study how early life stress (ELS) affects the ability to learn to feel calm.

Objective:

- To see if people with alcohol dependence and/or ELS have a harder time learning to feel calm than people without these. Also, to see if DNA is changed by ELS and if this change affects fear conditioning and extinction.

Eligibility:

* Adults ages 21-65 with and without an alcohol use disorder (AUD) and with and without ELS.
* Healthy volunteers.

Design:

* Participants will be screened with:

  * Medical history
  * Physical exam
  * Blood and urine tests
  * Psychological tests
  * Treatment for symptoms of alcohol withdrawal, if needed
* Healthy volunteers will have 1 overnight visit (2 days, 1 night). AUD participants will stay at the clinic for about 4 weeks.
* Participants will:

  * Rate alcohol use/craving, depression, anxiety, and childhood trauma.
  * Have psychophysiological measures: electrodes and mild electric shock.
* Have a functional magnetic resonance imaging (MRI) scan. Participants will lie on a table in a metal cylinder with a coil over their head. In the first scanning session, they will see pictures, do a simple task, and may get shocks. Participants will also do a second scanning session in which they will perform the aforementioned fear conditioning and extinction task, as well as a facial expression matching task, an affective word processing task, and a task measuring valuation of monetary rewards.

  * Answer questions about their emotions (some participants).
  * Have blood drawn from an arm vein or intravenous (IV) line.
  * AUD participants will get a dexamethasone pill. The next day, they will get a hormone injected in and have blood drawn from an IV line.
* AUD participants will have 3 follow-up visits with questions and blood and lab tests.

DETAILED DESCRIPTION:
Objective:

The primary goal of this study is to evaluate the role and interaction of (epi)genetic factors, early life stress (ELS) exposure, and alcohol use disorder (AUD) on neuronal mechanisms of fear conditioning and extinction.

The central hypothesis is that participants with AUD and ELS will have disrupted fear extinction, and in addition, those with ELS will also have disrupted fear extinction. AUD with ELS will have the most severe disruption of fear extinction as observed clinically in alcoholics with severe trauma - often presenting with the most severe phenotypes and being most treatment resistant. A disruption in fear extinction or living in constant fear after stress/trauma could thus put the individual at risk for AUD.

Identification and characterization of the neurobiological correlates underlying this mechanism is thus essential and could provide new avenues for treatment of AUD; namely developing interventions that normalize abnormal fear extinctions. These interventions could be for example, cognitive-behavior based or molecular by targeting genetic/epigenetic pathways potentially identified.

Our proposal, if successful, will first establish a reliable measureable endophenotype of fear extinction in AUD/ELS, both behaviorally (skin conductance response) and neuronal (using an fMRI paradigm). Furthermore, we will carry out exploratory genetic and epigenetics studies that might influence these measures. This model can then be used in follow up studies for novel therapeutic interventions that could target treatment of these mechanisms in AUD.

Study Population:

The study sample includes two patient groups and two control groups:

1. treatment-seeking or non-treatment-seeking individuals with AUD and ELS exposure;
2. treatment-seeking or non-treatment-seeking individuals with AUD without ELS exposure;
3. healthy volunteers with ELS exposure;
4. healthy volunteers without ELS exposure.

Target accrual for each of these groups is 25.

Design:

Subjects will be evaluated for fear conditioning and extinction using shock conditioning (extinction procedure combined with fMRI imaging that utilizes galvanic skin response). All participants will undergo whole-genome methylome analyses to assess genome wide methylation patterns. Genotyping of variants in candidate genes implicated in the biology of fear conditioning/extinction will be carried out.

Outcome Parameters:

The primary outcome of interest is fear extinction, measured by fMRI paradigms. Secondary objectives include: (1) explore the role of genetic variants and epigenetic factors and their impact on fear extinction in AUD and healthy controls with or without ELS; (2) explore differences in reward processing and emotion processing, measured by fMRI as a function of AUD, ELS, and (epi)genetic modulators; and (3) examine the relationship between fear extinction and clinical outcomes in both AUD and ELS participants sample.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Inclusion and exclusion criteria will be evaluated following screening conducted under the NIAAA screening protocols (98-AA-009 and/or 14-AA-0181).

INCLUSION CRITERIA:

INCLUSION CRITERIA FOR AUD GROUP:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding, agree to abstain or use accepted form of contraception
* Diagnosed with current alcohol dependence according to Diagnostic and Statistical Manual for Mental Disorders-Fourth Edition (DSM IV)
* Alcohol consumption within the past month provided by self-report
* Specify alcohol as their preferred drug in a clinical interview
* 98-AA-0009 and/or 14-AA-0181 screening consents signed
* Cleared venous access assessment
* Additional inclusion criteria for non-treatment seeking AUD: Able and willing to abstain from consuming alcohol 1 day prior to each study visit

INCLUSION CRITERIA FOR NON-AUD (HEALTHY VOLUNTEER) GROUP:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding, agree to abstain or use accepted form of contraception
* 98-AA-0009 and/or 14-AA-0181 screening consents signed
* Cleared venous access assessment

EXCLUSION CRITERIA:

EXCLUSION CRITERIA FOR AUD GROUP:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed, but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or current substance dependence other than alcohol, nicotine, or caffeine.
* Major medical problems (e.g., central nervous system (CNS), cardiovascular, respiratory, gastrointestinal (GI), hepatic, renal, endocrine, HIV, reproductive) that in the judgment of the PI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center.
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report
* Left-handedness
* Use of intrauterine device (IUD)
* Excluded from the optional DEX-CRH test if:

  * Allergy to dexamethasone or CRH
  * Use of medications that can affect the results of the test, including certain antibiotics, anti-seizure drugs, corticosteroids, and hormonal contraception
* Additional exclusionary criteria for non-treatment seeking AUD:

  * Presence of significant alcohol withdrawal symptoms, defined as a CIWA-Ar > 8.
  * History of epilepsy or alcohol-related seizures.
  * Are currently seeking treatment for alcohol problems

EXCLUSION CRITERIA FOR NON-AUD (HEALTHY VOLUNTEER) GROUP:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam.
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed, but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or substance dependence other than nicotine, or caffeine.
* Major medical problems (e.g., CNS, cardiovascular, respiratory, GI, hepatic, renal, endocrine, HIV, reproductive) that in the judgment of the PI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report
* Current or past DSM IV diagnosis of alcohol dependence or abuse
* Currently seeking treatment for alcohol problems as assessed by self-report
* Positive urine drug test at screening (for opiates, cannabinoids, amphetamines, cocaine, benzodiazepines)
* Positive breathalyzer test at screening
* Alcohol abstainer (never consumed alcohol in entire life)
* Left-handedness
* Use of intrauterine device (IUD)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AUD participants will be recruited from participants in the NIAAA screening platform protocols 14-AA-0181. Non-AUD participants will be recruited from participants in the NIAAA protocol 14-AA-0181. We will recruit all racial and ethnic groups in the greater Washington DC area
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the role and interaction of epigenetic/genetic factors, ELS exposure, and AUD on neuronal mechanisms of fear conditioning and extinction. | ongoing
  1) Fear extinction (extinction learning) is disrupted in AUD and differs between normal controls with or without ELS and AUD with or without ELS as measured by behavior (skin conductance response) and by fMRI (region of interest BOLD activation). 1a) AUD with ELS will have more severe disruption in their extinction learning phenotype. 2) Neuronal mechanisms involved in abnormal fear extinction in AUD include decreased vmPFC activation during fear which results in impaired inhibitory top-down control of the amygdala by the mPFC resulting in anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Falk W Lohoff, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grant BF, Stinson FS, Dawson DA, Chou SP, Dufour MC, Compton W, Pickering RP, Kaplan K. Prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2004 Aug;61(8):807-16. doi: 10.1001/archpsyc.61.8.807. PMID 15289279
- [Background] Heilig M, Thorsell A, Sommer WH, Hansson AC, Ramchandani VA, George DT, Hommer D, Barr CS. Translating the neuroscience of alcoholism into clinical treatments: from blocking the buzz to curing the blues. Neurosci Biobehav Rev. 2010 Nov;35(2):334-44. doi: 10.1016/j.neubiorev.2009.11.018. Epub 2009 Nov 24. PMID 19941895
- [Background] Goldman D, Oroszi G, Ducci F. The genetics of addictions: uncovering the genes. Nat Rev Genet. 2005 Jul;6(7):521-32. doi: 10.1038/nrg1635. PMID 15995696
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AA-0127.html